CLINICAL TRIAL: NCT03789396
Title: Pilot Study of Targeted Normoxia in Critically Ill Trauma Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 18-1528
Record Dates: First submitted 2018-12-13; First posted 2018-12-28 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-06

CONDITIONS: Trauma; Critical Illness; Oxygen Toxicity
Keywords: Oxygenation; Hypoxia; Normoxia; Hyperoxia; Trauma; Critical Illness
MeSH Terms: conditions — Wounds and Injuries; Critical Illness; Hypoxia; Hyperoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation: The control groups will be trauma patients admitted to the ICU 12 months prior to targeted normoxia
  Interventions: Other: Usual Care Oxygenation
- Post-implementation: The intervention group will be trauma patients admitted to the ICU during the 6 months after the targeted normoxia implementation.
  Interventions: Other: Targeted Normoxia (oxygen saturation 90-96%)

INTERVENTIONS:
Other: Targeted Normoxia (oxygen saturation 90-96%) — The intervention (post-implementation) group will be trauma patients admitted to the ICU during the 6 months after the targeted normoxia implementation
  Groups: Post-implementation
Other: Usual Care Oxygenation — The control (pre-implementation) group will be trauma patients admitted to the ICU during the 12 months prior to the targeted normoxia implementation
  Groups: Pre-implementation

SUMMARY:
The objective of this study is to conduct an observational pre/post study to evaluate the clinical impact oxygen guideline implementation on oxygen utilization and oxygenation in critically ill trauma patients.

DETAILED DESCRIPTION:
Supplemental oxygen is fundamental in caring for critically ill trauma. While the avoidance of hypoxia is vital, the current clinical practice of excessive oxygenation settings is common, and unnecessary, and may even be harmful.

An expert panel convened to define optimal oxygenation targets in critically ill trauma patients. The strong consensus was to target normoxia at an oxygen saturation (SpO2) range of 90-96% and arterial oxygen (PaO2) range of 60-100 mmHg. Accordingly, a pilot trial implementation of this consensus will occur for the care of trauma patients.

Specific Aim:

This is an observational pre/post study to evaluate the impact of targeted normoxia implementation in optimizing oxygen delivery and oxygenation in critically ill trauma patients.

Hypotheses:

That the clinical efforts to improve adherence to oxygen guidelines will:

1. improve the proportion of time spent with target normoxia thresholds (oxygen saturation SpO2 90-96%) by
2. reducing utilization of unnecessary supplementation oxygen
3. without a substantive increase in hypoxic episodes or an adverse impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Acute Injury/Trauma
* Arrival to Emergency Department

Exclusion Criteria:

* <18 years of age
* Known prisoners

Ages: 18 Years to 109 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adit Ginde, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuroda N, Tsutsumi Y, Banno M. Does statistical difference in the pre/post-quasi-experimental study mean the utility of multimodal educational intervention in targeted normoxia in critically ill trauma patients? J Trauma Acute Care Surg. 2021 Aug 1;91(2S Suppl 2):S269-S270. doi: 10.1097/TA.0000000000003301. No abstract available. PMID 34039929

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-implementation | Post-implementation
Started | 371 | 201
Completed | 371 | 201
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-implementation: The control groups will be trauma patients admitted to the ICU 12 months prior to targeted normoxia (admitted January 1, 201 to December 31, 2018).
  Usual Care Oxygenation: The control (pre-implementation) group will be trauma patients admitted to the ICU during the 12 months prior to the targeted normoxia implementation
- Post-implementation: The intervention group will be trauma patients admitted to the ICU during the 6 months after the targeted normoxia implementation (admitted January 1, 2019+ to July 1, 2019).
  Targeted Normoxia (oxygen saturation 90-96%): The intervention (post-implementation) group will be trauma patients admitted to the ICU during the 6 months after the targeted normoxia implementation
- Total: Total of all reporting groups
Arm/Group | Pre-implementation | Post-implementation | Total
Number analyzed (Participants) | 371 | 201 | 572
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (21.4) | 52.5 (21.4) | 54.3 (21.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 62 | 175
  Male | 258 | 139 | 397
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 51 | 134
  Not Hispanic or Latino | 243 | 134 | 377
  Unknown or Not Reported | 45 | 16 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 20 | 69
  White | 194 | 114 | 308
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 128 | 67 | 195

OUTCOME MEASURES:

1. Primary Outcome: Patient-time Hyperoxic and Not on Room Air
Description: Total percentage of patient-time hyperoxic and not on room air: total time spent by patients in a hyperoxic state while receiving supplemental oxygen, divided by total patient time on study
Time Frame: From time of emergency department arrival until the date of hospital discharge or death, assessed up to 28 days from dates Jan. 1, 2018 to July 1, 2019
Measure: Mean (Standard Error); unit: Percent patient-time in hyperoxia
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Percent patient-time in hyperoxia | 40.6 (2.5) | 33.9 (3.3)
Statistical Analysis 1: Comparison: Pre-implementation vs Post-implementation; Comparison of patient odds of being hyperoxic and not on room air pre- versus post-intervention; Test type: Superiority; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.57 to 0.97], Standard Error of Mean 0.14

2. Secondary Outcome: Episodes of Hypoxia (SpO2< 88%)
Description: SpO2 saturations below 88%. Episodes of hypoxia reported in minutes (i.e. one episode of hypoxia = one minute spent).
Time Frame: From time of emergency department arrival until the date of hospital discharge or death, assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Minutes | 12 [0 to 75] | 14 [0 to 70]

3. Secondary Outcome: Episodes of Hyperoxia (SpO2 >96%)
Description: SpO2 saturations above 96%. Episodes of hyperoxia reported in minutes (i.e. one episode of hyperoxia = one minute spent).
Time Frame: From time of emergency department arrival until the date of hospital discharge or death, assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Minutes | 3151 [1274 to 5559] | 3037 [1455 to 5010]

4. Secondary Outcome: Ventilator Free Day
Description: Ventilator Free Days = Days off ventilator
Time Frame: From time of emergency department arrival until the date of hospital discharge or death, assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Days | 28 [24 to 28] | 28 [24 to 28]

5. Secondary Outcome: Time to Room Air
Description: Duration of supplemental oxygen use measured in days
Time Frame: From time of emergency department arrival until the date of hospital discharge or death, assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Days | 2 [0 to 4] | 2 [1 to 4]

6. Secondary Outcome: Measured by Daily Sequential Organ Failure Assessment (SOFA)
Description: Acute organ injury as measured by SOFA score
Time Frame: First 7 days of hospitalization
Population: Variables necessary to determine SOFA could not be collected and, therefore, no analysis can be reported (cite: Dylla L, Anderson EL, Douin DJ, et al. A quasiexperimental study of targeted normoxia in critically ill trauma patients. J Trauma Acute Care Surg. 2021;91(2S Suppl 2):S169-S175.).
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: ICU Length of Stay
Description: Number of days spent in the ICU
Time Frame: From time of emergency department arrival until the date of ICU discharge or death, assessed up to 180 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Days | 10.9 (26.8) | 10.4 (14.0)

8. Secondary Outcome: Hospital Length of Stay
Description: Number of days spent in the hospital
Time Frame: From time of emergency department arrival until the date of hospital discharge or death, assessed up to 180 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Days | 6 [3 to 13] | 7 [4 to 15]

9. Secondary Outcome: Hospital Discharge Disposition
Description: Percent of patients discharged to home or facility vs death or hospice = measuring illness at discharge
Time Frame: Date of hospital discharge, assessed up to 180 days
Measure: Mean (Standard Error); unit: Percent of patients as described
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Percent of patients as described | 71.4 (2.3) | 71.1 (3.2)

10. Secondary Outcome: Hospital Mortality
Description: Percent of deceased participants
Time Frame: From time of emergency department arrival until the date of hospital discharge or death, assessed up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 371 | 201
Participants | 21 | 16

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Pre-implementation | Post-implementation
All-Cause Mortality (participants affected / at risk) | 0/371 | 0/201
Serious Adverse Events (participants affected / at risk) | 0/371 | 0/201
Other Adverse Events (participants affected / at risk) | 0/371 | 0/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT03789396/Prot_SAP_000.pdf